CLINICAL TRIAL: NCT06301516
Title: Impact Virtual Reality: An Emotion Recognition and Regulation Training Program for Youth With Conduct Disorder
Brief Title: Impact VR: An Emotion Recognition and Regulation Training Program for Youth With CD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20027823; R41MH133540 (NIH)
Record Dates: First submitted 2024-02-19; First posted 2024-03-08 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Conduct Disorder; Conduct Disorders in Children; Conduct Disorders in Adolescence; Callous-Unemotional Traits
Keywords: Conduct Problems
MeSH Terms: conditions — Conduct Disorder

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial of psychological intervention. Once all assessments are completed, the treatment group allocation will be disclosed to the administrating researcher, youth, and caregiver. This blinded approach to block randomization prevents any bias from occurring during the assessment phase by the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Impact VR (Experimental): Participants enrolled into Impact VR will be complete the first of four sessions. The four 20-minute sessions will be completed over 4 weeks (one session per week) either in the lab, at the participant's home, school or a mutual private meeting place
  Interventions: Behavioral: Virtual Reality
- Comparative Control (Other): Participants enrolled into the comparative control group will complete a one-time PowerPoint presentation that provides an overview of emotion expressions and instructions on how to recognize emotions in others
  Interventions: Other: Comparative Control

INTERVENTIONS:
Behavioral: Virtual Reality — VR: The goal of the VR intervention is to provide youth an immersive, engaging, and therapeutic environment to reduce CD and CU traits
  Arms: Experimental: Impact VR
Other: Comparative Control — Complete a one-time PowerPoint presentation that provides an overview of emotion expressions and instructions on how to recognize emotions in others.
  Arms: Comparative Control

SUMMARY:
Conduct disorder (CD) is one of the most prevalent childhood psychiatric disorders. Unfortunately, there are limited treatments available for CD. The present study aims to test an innovative virtual reality intervention called Impact VR for symptom reduction in a sample of 60 youth with CD.

DETAILED DESCRIPTION:
Within the CD diagnosis, a subset of youth (12-46%) display callous-unemotional (CU) traits (termed "limited prosocial emotions"). CU traits denote additional symptoms including a lack of remorse/guilt, a callous lack of empathy, shallow affect, and/or lack of concern about performance. Although both CD and CU traits are inextricably linked to poor outcomes for youth, there remains a scarcity of targeted interventions for CD and CU traits. One of the most significant challenges for treatment is that youth with CD are often perceived by providers as treatment-resistant and treatment disrupters. This leads to poor treatment retention and further isolation from treatment opportunities. Further, existing interventions that target antisocial behaviors more generally are costly because they require 24/7 behavioral management therapies. Impact VR is a psychoeducational intervention for improving emotion recognition and regulation, using immersive gameplay and storylines that are relevant to youth. Impact VR uses evidence-based cognitive and dialectical behavioral approaches to improve emotion regulation. At the center of Impact VR is an individualized training program that teaches youth to effectively identify emotional expressions in others.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10-17 years old
* Identified through the TriNetX database as having a conduct disorder diagnosis
* English speaking

Exclusion Criteria:

* Youth aged <10 years and >18 years old
* Non-English speaking
* Youth of caregivers younger than 18 years old.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Assess the preliminary efficacy of Impact Virtual Reality (VR) in reducing Callous-Unemotional traits | Baseline, 1-month and 3-months post-randomization
  Participants enrolled into Impact VR will be complete the first of four sessions. The four 20-minute Callous-unemotional traits will be measured using the 24-item Inventory of Callous-Unemotional Traits. Both the parent and youth reports will be completed. sessions will be completed over 4 weeks (one session per week) either in the lab, at the participant's home, school or a mutual private meeting place.
Assess the preliminary efficacy of Impact Virtual Reality (VR) in reducing Conduct disorder | Baseline, 1-month and 3-months post-randomization
  Conduct disorder symptoms will be measured using the Kiddie Schedule for Affective Disorders and Schizophrenia, which is a semi-structured interview administered to the caregiver and child.
Assess the preliminary efficacy of Impact Virtual Reality (VR) in reducing Conduct Problems | Baseline, 1-month and 3-months post-randomization
  Conduct problems will be assessed using parent and child reports on the Behavior Assessment System for Children, 3rd edition (BASC-3)
Assess the preliminary efficacy of Impact Virtual Reality (VR) in reducing Emotion regulation | Baseline, 1-month and 3-months post-randomization
  Emotion Regulation will be assessed using parent and child reports on the Behavior Assessment System for Children, 3rd edition (BASC-3).
Assess the preliminary efficacy of Impact Virtual Reality (VR) in reducing Emotion recognition | Baseline, 1-month and 3-months post-randomization
  Emotion recognition will be measured using the Penn Emotion Recognition Test, which is a computer-based task completed by the youth

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Thomson, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT06301516/Prot_000.pdf